CLINICAL TRIAL: NCT02929875
Title: Assessing the Effect of Education Based on Theory of Planned Behavior (TPB) on Delivery Type Selection in Pregnant Women Referring to Kermanshah Health Centers at 1393
Brief Title: The Effect of Educational Intervention on Delivery Type Selection in Pregnant Women at Kermanshah, Iran
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ilam University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zeinab Ghazanfari, Academic member, Ilam University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 944012/99
Record Dates: First submitted 2016-10-08; First posted 2016-10-11 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case (Educational based on TPB) (Experimental): Educational intervention delivered to subjects. The content of education includes:
  Three training sessions were given to the case group; each lasted for one hour, during a period of twenty days. During each one-hour training session a period of 45 minutes was dedicated to listening to lectures, having discussions, and discussing methods of using teaching aids such as pamphlets and manuals. The last 15 minutes was used to summarize issues and answer questions.
  Interventions: Behavioral: Education based on TPB
- Control (No intervention) (No Intervention): No educational intervention provided to subjects in control group

INTERVENTIONS:
Behavioral: Education based on TPB — Three Training sessions were given to the case group; each lasted for one hour, during a period of twenty days. During each one-hour training session a period of 45 minutes was dedicated to listening to lectures, having discussions, and discussing methods of using teaching aids such as pamphlets and manuals. The last 15 minutes was used to summarize issues and answer questions.
  Arms: Case (Educational based on TPB)

SUMMARY:
In an experimental research, 100 nulliparous pregnant women who had referred to health care centers in Kermanshah were randomly selected and after taking Written Informed Consent letter, assigned into case and control groups. instruction based on TPB was provided just for the case group. Afterwards, post-test was taken by both groups and the results were analyzed.

DETAILED DESCRIPTION:
In an experimental research, 100 nulliparous pregnant women with the gestational age of 28-36 weeks who had referred to health care centers in Kermanshah (western Iran) were randomly selected and after taking Written Informed Consent letter, assigned into case and control groups. The inclusion criteria consisted of nulliparous pregnant women with the gestational age of 28-36 weeks, women under 35 years old, and no contraindications for normal childbirth. Exclusion criteria included the absence of women in continuous training sessions, premature delivery, and maternal unavailability during the completion of the questionnaires.

Three Training sessions each lasted for one hour during twenty days were hold for the case group. The first session was conducted to affect their attitude and provide favourable attitude towards natural delivery. The second session was allocated to presenting feasible methods for reducing pain in order to enhance mothers' perceived behavioral control. In the 3rd session the methods were exercised practically so that they could better employ them whenever needed during the parturition. As a result, the mothers' selection of the sort of delivery was checked out. In order to influence the subjective norm, pregnant women were also asked to transfer their knowledge to their husbands. The control group also received only routine training sessions by the midwives in the health care centers.

In each one-hour training session; 45 minutes was dedicated to listening to lectures, having colloquies, and discussing methods via using teaching aids such as pamphlets, and manuals. The last 15 minutes was allocated to summarizing the issues and answering mothers' questions.

At the end of the training sessions, the post-test was administered for both groups and the data were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* consisted of nulliparous pregnant women with the gestational age of 28-36 weeks, women under 35 years old, informed consent of the mother and her husband, and no contraindications for normal childbirth.

Exclusion Criteria:

* Included the absence of women in continuous training sessions, premature delivery, and maternal unavailability during the completion of the questionnaires.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
frequency of child birth by Vaginal/Natural Delivery method. | 3 Months
  such data are registered officially in hospitals and health centers. we collect the data through seeing the documents

IPD SHARING:
Plan to Share IPD: No